CLINICAL TRIAL: NCT00637910
Title: Optimization of Erlotinib for the Treatment of Patients With Advanced Non Small Cell Lung Cancer: an Italian Randomized Trial
Brief Title: Tarceva Italian Lung Optimization tRial
Acronym: TAILOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatebenefratelli and Ophthalmic Hospital (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Niguarda Hospital (Other)
Responsible Party: Principal Investigator, Scanni Alberto, Alberto Scanni MD, Fatebenefratelli and Ophthalmic Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM6F5JER; 2007-004786-17 (EudraCT Number)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Advanced NSCLC; EGFR; EGFR copy number; Kras mutations; EGRF mutations; Docetaxel; Erlotinib; Polymorphisms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib Arm (Experimental)
  Interventions: Drug: Erlotinib
- Docetaxel Arm (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg/day per os until disease progression or unacceptable toxicity develops
  Other Names: Tarceva
  Arms: Erlotinib Arm
Drug: Docetaxel — Docetaxel 75 mg/mq on day 1, every 21 days (3-weekly schedule) or Docetaxel 35 mg/mq 0n day 1,8 and 15 every 28 days (weekly schedule). _Until disease progression or unacceptable toxicity develops
  Other Names: Taxotere
  Arms: Docetaxel Arm

SUMMARY:
The aim of this study is to assess the superiority of docetaxel in comparison to erlotinib in second line in wild-type EGFR tumour patients.

DETAILED DESCRIPTION:
Erlotinib is registered in all patients affected with NSCLC in second and subsequent lines with a small benefit on Overall Survival. Recent evidence suggest that patients with EGFR mutations have a clear benefit when they are treated with EGFR tyrosine kinase inhibitors, while the role of these drugs in wild-type EGFR patients, that are representing the large majority (about 85-90%), is still unclear and no properly planned trials assessed before this issue. Recently, indirect evidence on subgroup analyses on randomized trial suggest that chemotherapy might be superior to erlotinib in wild-type EGFR patients.

Moreover, several authors do not recommend the use of EGFR determined with immunohistochemistry (IHC) or FISH because they do not reproducibly predict outcome.

For these reasons the protocol was amended in May 2011 in a superiority trial of docetaxel versus erlotinib, while the first version was aimed to assess the interaction with biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histological or cytological confirmation of NSCLC (may be from initial diagnosis of NSCLC or subsequent biopsy). Only patients with available tissue samples may be included in the study
* Absence of EGFR mutations of exons 19 or 21 (randomization)
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy
* One prior platinum-based at adequate doses and taxane free regimen
* Measurable (uni-dimensional) disease by RECIST in a lesion not previously irradiated or non-measurable disease
* ECOG-PS 0-2
* ANC greater than 1.5 x 109/L and platelets greater than 100 x 109/L
* Bilirubin level either normal or <1.5xULN
* AST (SGOT) and ALT (SGPT) <2.5xULN (≤5 x ULN if liver metastases are present)
* Serum creatinine <1.5xULN
* Effective contraception for both, male and female pts, if the risk of conception exists
* Recovery from all acute toxicities of prior therapies
* Provision of written informed consent to the analysis of biological markers (registration)
* Provision of written informed consent to enter the randomized part of the study (randomization)

Exclusion Criteria:

* Prior therapy with an experimental agent whose primary mechanism of action is inhibition of EGFR or its associated tyrosine kinase
* Prior chemotherapy with taxanes
* Newly diagnosed CNS metastases that have not yet been treated with surgery and/or radiation. Pts with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically SD (no steroid therapy or steroid dose being tapered) for at least 28 daysLess than 14 days since completion of prior radiotherapy or persistence of any radiotherapy related toxicity
* Any unresolved chronic toxicity from previous anticancer therapy that, in the opinion of the investigator, makes it inappropriate for the patient to be enrolled in the study Known severe hypersensitivity to erlotinib or any of the excipients of this product
* Known hypersensitivity to docetaxel, polysorbate 80 or other drugs formulated with polysorbate 80, or any of the excipients of docetaxel
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Unable to swallow tablets
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic or patients with uncomplicated progressive lymphangitic carcinomatosis need not be excluded)
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* As judged by the investigator, any inflammatory changes of the surface of the eye
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2007-11; Primary Completion 2012-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 12 months after the last patient is randomized

SECONDARY OUTCOMES:
Progression Free Survival | with 4 years and 12 months after the last patient is randomized
Response assessed with RECIST criteria | within 4 years
Quality of Life assessed with QLQ-C30 and QLQ-LC13 questionnaires | within 4 years
Toxicity, graded according to the NCI-CTAE version 3.0 | within 4 years
Frequency and nature of serious adverse reactions | within 4 years
Premature withdrawals | within 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Scanni, MD, Principal Investigator — Fatebenefratelli and Ophthalmic Hospital
Locations (104):
- Italy (104):
  - S. Giovanni di Dio Hospital, Agrigento, Agrigento
  - Ospedale Civili Riuniti Giovanni Paolo II, Sciacca, Agrigento
  - Fabriano Hospital, Fabriano, Ancona
  - Ospedali Riuniti Umberto I - Lancisi - Salesi, Torrette, Ancona
  - Oncologia A.S.L. AV1, Ariano Irpino, Avellino
  - Azienda Ospedaliera Universitaria Consorziale Policlinico, Bari, Bari
  - Fatebenefratelli Hospital, Benevento, Benevento
  - G. Rummo Hospital, Benevento, Benevento
  - Pesenti-Fenaroli Hospital, Alzano Lombardo, Bergamo
  - Ospedali Riuniti, Bergamo, Bergamo
  - Ospedale di Vipiteno, Sterzing, Bolzano
  - Oncologia Medica Azienda Spedali Civili, Brescia, BS
  - Pneumologia Azienda Spedali Civili, Brescia, BS
  - Ospedale centrale di Bolzano, Bolzano, BZ
  - Armando Businco Oncological Hospital, Cagliari, Cagliari
  - Policlinico Universitario di Monserrato, Monserrato, Cagliari
  - Presidio Ospedaliero Cardarelli ASL 3, Campobasso, Campobasso
  - Ospedale Santa Barbara, Iglesias, Carbonia Iglesias
  - Renzetti Hospital, Lanciano, Chieti
  - Ospedale S. Elia, Caltanissetta, CL
  - Sant'Anna Hospital, Como, Como
  - Mariano Santo Hospital, Cosenza, Cosenza
  - San Francesco Hospital, Paola, Cosenza
  - Ospedale Maggiore di Crema, Crema, Crema
  - S. Croce e Carle Hospital, Cuneo, Cuneo
  - Ospedale Civile di Saluzzo Savigliano, Saluzzo, Cuneo
  - Istituto Toscano Tumori Ospedale S. Giuseppe Antica Sede, Empoli, Firenze
  - Azienda Ospedaliero Universitaria Careggi, Florence, Firenze
  - Galliera Hospital, Genova, Genova
  - Monfalcone Hospital, Monfalcone, Gorizia
  - F. Veneziale Hospital, Isernia, Isernia
  - Ospedale Civile Ferrari, Casarano, Lecce
  - Azienda Ospedaliera di Lecco, Lecco, Lecco
  - Ospedale Civile di Casalpusterlengo, Casalpusterlengo, Lodi
  - Ospedale S. Maria Goretti, Latina, LT
  - B. Eustachio Hospital, San Severino Marche, Macerata
  - San Vincenzo Hospital, Taormina, Messina
  - Azienda Ospedaliera Melegnano- P.O. Gorgonzola, Gorgonzola, Milano
  - Legnano Hospital, Legnano, Milano
  - Ospedale Civile di Legnano -Presidio di Magenta, Magenta, Milano
  - Fatebenefratelli and Ophthalmic Hospital, Milan, Milano
  - Fondazione Ospedale Maggiore Policlinico - Mangiagalli e Regina Elena, Milan, Milano
  - San Paolo Hospital, Milan, Milano
  - San Carlo Borromeo Hospital, Milan, Milano
  - Azienda Ospedaliera Luigi Sacco Polo Universitario, Milan, Milano
  - San Gerardo Hospital, Monza, Milano
  - Rho Hospital - Azienda Ospedaliera Salvini-Garbagnate, Rho, Milano
  - Policlinico San Donato, San Donato Milanese, Milano
  - IRCCS Multimedica, Sesto San Giovanni, Milano
  - Ospedale Civile di Vimercate, Vimercate, Milano
  - Vizzolo Predabissi Hospital, Vizzolo Predabissi, Milano
  - San Leonardo Hospital, Gragnano, Napoli
  - Cardarelli Hospital, Napoli, Napoli
  - D. Cotugno Hospital, Napoli, Napoli
  - San Gennaro Hospital - ASL NA 1, Napoli, Napoli
  - Ospedale Maggiore della Carità, Novara, Novara
  - Azienda Ospedaliera Universitaria Presidio "Paolo Giaccone", Palermo, Palermo
  - Presidio Ospedaliero "M. Ascoli" ARNAS Civico, Palermo, Palermo
  - Centro Oncologico "La Maddalena", Palermo, Palermo
  - Ospedale Civile Vigevano, Vigevano, Pavia
  - Policlinico Universitario Palermo, Palermo, PA
  - S. Maria della Misericordia Hospital, Perugia, Perugia
  - San Massimo Hospital, Penne, Pescara
  - Piacenza Hospital, Piacenza, Piacenza
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - S. Maria degli Angeli Hospital, Pordenone, Pordenone
  - Umberto I Hospital, Lugo, Ravenna
  - Ospedale Civile di Siderno - ASL n°9 Locri, Siderno, Reggio Calabria
  - S. Sebastiano Hospital, Correggio, Reggio Emilia
  - Arcispedale S. Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale di Scandiano, Scandiano, Reggio Emilia
  - Pneumologia Oncologica II-San Camillo Forlanini Hospital, Roma, Roma
  - Oncologia Medica-San Camillo Forlanini Hopsital, Roma, Roma
  - Università Campus Bio-Medico, Roma, Roma
  - Policlinico Umberto I, Roma, Roma
  - S. Giovanni - Addolorata Hospital, Roma, Roma
  - S. Giovanni Evangelista Hospital, Tivoli, Roma
  - ASL SA1 -P.O. Umberto I, Nocera Inferiore, Salerno
  - Azienda Ospedaliera S. Giovanni di Dio e Ruggi d'Aragona, Salerno, Salerno
  - Presidio Ospedaliero San Luca, Vallo della Lucania, Salerno
  - Ospedale Civile SS. Annunziata, Sassari, Sassari
  - Ospedale Valdichiana "Nottola", Montepulciano, Siena
  - Ospedale Valdelsa "Campostaggia", Poggibonsi, Siena
  - Sondrio Hospital-Azienda Ospedaliera Valtellina e Valchiavenna, Sondrio, Sondrio
  - Ospedale di Terni, Terni, TR
  - Multimedia Santa Maria, Castellanza, Varese
  - Azienda Ospedaliera Busto Arsizio, Saronno, Varese
  - Ospedale di Circolo, Varese, Varese
  - Umberto I Hospital, Mestre, Venezia
  - SS. Giovanni e Paolo Hospital, Venezia, Venezia
  - Ospedale Mater Salutis, Legnago, Verona
  - San Bartolo Hospital, Vicenza, Vicenza
  - Belcolle Hospital, Viterbo, Viterbo
  - Ospedale Policlinico G.B. Rossi, Verona, VR
  - Ospedale San Donato, Arezzo
  - A.O.U. S. Anna, Ferrara
  - A.O.U. Careggi, Florence
  - A.O. San Martino, Genova
  - A.O. Monaldi, Napoli
  - Ospedale Civile Santa Maria delle Croci, Ravenna
  - Ospedale San Pietro Fatebenefratelli, Roma
  - Universita' di Sassari Oncologia Medica, Sassari
  - Ospedale Morelli, Sondrio
  - A.O.U. San Giovanni Battista Molinette, Torino

REFERENCES:
- [Background] Greenlee RT, Hill-Harmon MB, Murray T, Thun M. Cancer statistics, 2001. CA Cancer J Clin. 2001 Jan-Feb;51(1):15-36. doi: 10.3322/canjclin.51.1.15. PMID 11577478
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Shepherd FA, Dancey J, Ramlau R, Mattson K, Gralla R, O'Rourke M, Levitan N, Gressot L, Vincent M, Burkes R, Coughlin S, Kim Y, Berille J. Prospective randomized trial of docetaxel versus best supportive care in patients with non-small-cell lung cancer previously treated with platinum-based chemotherapy. J Clin Oncol. 2000 May;18(10):2095-103. doi: 10.1200/JCO.2000.18.10.2095. PMID 10811675
- [Background] Schuette W, Nagel S, Blankenburg T, Lautenschlaeger C, Hans K, Schmidt EW, Dittrich I, Schweisfurth H, von Weikersthal LF, Raghavachar A, Reissig A, Serke M. Phase III study of second-line chemotherapy for advanced non-small-cell lung cancer with weekly compared with 3-weekly docetaxel. J Clin Oncol. 2005 Nov 20;23(33):8389-95. doi: 10.1200/JCO.2005.02.3739. PMID 16293869
- [Background] Hanna N, Shepherd FA, Fossella FV, Pereira JR, De Marinis F, von Pawel J, Gatzemeier U, Tsao TC, Pless M, Muller T, Lim HL, Desch C, Szondy K, Gervais R, Shaharyar, Manegold C, Paul S, Paoletti P, Einhorn L, Bunn PA Jr. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004 May 1;22(9):1589-97. doi: 10.1200/JCO.2004.08.163. PMID 15117980
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Herbst RS, Prager D, Hermann R, Fehrenbacher L, Johnson BE, Sandler A, Kris MG, Tran HT, Klein P, Li X, Ramies D, Johnson DH, Miller VA; TRIBUTE Investigator Group. TRIBUTE: a phase III trial of erlotinib hydrochloride (OSI-774) combined with carboplatin and paclitaxel chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5892-9. doi: 10.1200/JCO.2005.02.840. Epub 2005 Jul 25. PMID 16043829
- [Background] Gatzemeier U, Pluzanska A, Szczesna A, Kaukel E, Roubec J, De Rosa F, Milanowski J, Karnicka-Mlodkowski H, Pesek M, Serwatowski P, Ramlau R, Janaskova T, Vansteenkiste J, Strausz J, Manikhas GM, Von Pawel J. Phase III study of erlotinib in combination with cisplatin and gemcitabine in advanced non-small-cell lung cancer: the Tarceva Lung Cancer Investigation Trial. J Clin Oncol. 2007 Apr 20;25(12):1545-52. doi: 10.1200/JCO.2005.05.1474. PMID 17442998
- [Background] Marchetti A, Martella C, Felicioni L, Barassi F, Salvatore S, Chella A, Camplese PP, Iarussi T, Mucilli F, Mezzetti A, Cuccurullo F, Sacco R, Buttitta F. EGFR mutations in non-small-cell lung cancer: analysis of a large series of cases and development of a rapid and sensitive method for diagnostic screening with potential implications on pharmacologic treatment. J Clin Oncol. 2005 Feb 1;23(4):857-65. doi: 10.1200/JCO.2005.08.043. PMID 15681531
- [Background] Sequist LV, Joshi VA, Janne PA, Muzikansky A, Fidias P, Meyerson M, Haber DA, Kucherlapati R, Johnson BE, Lynch TJ. Response to treatment and survival of patients with non-small cell lung cancer undergoing somatic EGFR mutation testing. Oncologist. 2007 Jan;12(1):90-8. doi: 10.1634/theoncologist.12-1-90. PMID 17285735
- [Background] Taron M, Ichinose Y, Rosell R, Mok T, Massuti B, Zamora L, Mate JL, Manegold C, Ono M, Queralt C, Jahan T, Sanchez JJ, Sanchez-Ronco M, Hsue V, Jablons D, Sanchez JM, Moran T. Activating mutations in the tyrosine kinase domain of the epidermal growth factor receptor are associated with improved survival in gefitinib-treated chemorefractory lung adenocarcinomas. Clin Cancer Res. 2005 Aug 15;11(16):5878-85. doi: 10.1158/1078-0432.CCR-04-2618. PMID 16115929
- [Background] van Zandwijk N, Mathy A, Boerrigter L, Ruijter H, Tielen I, de Jong D, Baas P, Burgers S, Nederlof P. EGFR and KRAS mutations as criteria for treatment with tyrosine kinase inhibitors: retro- and prospective observations in non-small-cell lung cancer. Ann Oncol. 2007 Jan;18(1):99-103. doi: 10.1093/annonc/mdl323. Epub 2006 Oct 23. PMID 17060486
- [Background] Cappuzzo F, Hirsch FR, Rossi E, Bartolini S, Ceresoli GL, Bemis L, Haney J, Witta S, Danenberg K, Domenichini I, Ludovini V, Magrini E, Gregorc V, Doglioni C, Sidoni A, Tonato M, Franklin WA, Crino L, Bunn PA Jr, Varella-Garcia M. Epidermal growth factor receptor gene and protein and gefitinib sensitivity in non-small-cell lung cancer. J Natl Cancer Inst. 2005 May 4;97(9):643-55. doi: 10.1093/jnci/dji112. PMID 15870435
- [Background] Bell DW, Lynch TJ, Haserlat SM, Harris PL, Okimoto RA, Brannigan BW, Sgroi DC, Muir B, Riemenschneider MJ, Iacona RB, Krebs AD, Johnson DH, Giaccone G, Herbst RS, Manegold C, Fukuoka M, Kris MG, Baselga J, Ochs JS, Haber DA. Epidermal growth factor receptor mutations and gene amplification in non-small-cell lung cancer: molecular analysis of the IDEAL/INTACT gefitinib trials. J Clin Oncol. 2005 Nov 1;23(31):8081-92. doi: 10.1200/JCO.2005.02.7078. Epub 2005 Oct 3. PMID 16204011
- [Background] Hirsch FR, Varella-Garcia M, Bunn PA Jr, Franklin WA, Dziadziuszko R, Thatcher N, Chang A, Parikh P, Pereira JR, Ciuleanu T, von Pawel J, Watkins C, Flannery A, Ellison G, Donald E, Knight L, Parums D, Botwood N, Holloway B. Molecular predictors of outcome with gefitinib in a phase III placebo-controlled study in advanced non-small-cell lung cancer. J Clin Oncol. 2006 Nov 1;24(31):5034-42. doi: 10.1200/JCO.2006.06.3958. PMID 17075123
- [Background] Cappuzzo F, Varella-Garcia M, Shigematsu H, Domenichini I, Bartolini S, Ceresoli GL, Rossi E, Ludovini V, Gregorc V, Toschi L, Franklin WA, Crino L, Gazdar AF, Bunn PA Jr, Hirsch FR. Increased HER2 gene copy number is associated with response to gefitinib therapy in epidermal growth factor receptor-positive non-small-cell lung cancer patients. J Clin Oncol. 2005 Aug 1;23(22):5007-18. doi: 10.1200/JCO.2005.09.111. PMID 16051952
- [Background] Cappuzzo F, Magrini E, Ceresoli GL, Bartolini S, Rossi E, Ludovini V, Gregorc V, Ligorio C, Cancellieri A, Damiani S, Spreafico A, Paties CT, Lombardo L, Calandri C, Bellezza G, Tonato M, Crino L. Akt phosphorylation and gefitinib efficacy in patients with advanced non-small-cell lung cancer. J Natl Cancer Inst. 2004 Aug 4;96(15):1133-41. doi: 10.1093/jnci/djh217. PMID 15292385
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Bergman B, Aaronson NK, Ahmedzai S, Kaasa S, Sullivan M. The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials. EORTC Study Group on Quality of Life. Eur J Cancer. 1994;30A(5):635-42. doi: 10.1016/0959-8049(94)90535-5. PMID 8080679
- [Background] Osoba D, Bezjak A, Brundage M, Zee B, Tu D, Pater J; Quality of Life Committee of the NCIC CTG. Analysis and interpretation of health-related quality-of-life data from clinical trials: basic approach of The National Cancer Institute of Canada Clinical Trials Group. Eur J Cancer. 2005 Jan;41(2):280-7. doi: 10.1016/j.ejca.2004.10.017. PMID 15661554
- [Background] Armstrong BG, Sloan M. Ordinal regression models for epidemiologic data. Am J Epidemiol. 1989 Jan;129(1):191-204. doi: 10.1093/oxfordjournals.aje.a115109. PMID 2910061
- [Background] Crinò L; Zatloukal P; Reck M; Pesek M; Thomson J; Ford H; Hirsch F; Duffield E; Armour A; Cullen M. Gefitinib (Iressa) versus vinorelbine in chemonaive elderly pts with advanced NSCLC (INVITE): a randomized phase II study: B3-04. Journal of Thoracic Oncology Volume 2(8) Supplement 4 August 2007p S341 number 8
- [Background] Keedy VL, Temin S, Somerfield MR, Beasley MB, Johnson DH, McShane LM, Milton DT, Strawn JR, Wakelee HA, Giaccone G. American Society of Clinical Oncology provisional clinical opinion: epidermal growth factor receptor (EGFR) Mutation testing for patients with advanced non-small-cell lung cancer considering first-line EGFR tyrosine kinase inhibitor therapy. J Clin Oncol. 2011 May 20;29(15):2121-7. doi: 10.1200/JCO.2010.31.8923. Epub 2011 Apr 11. PMID 21482992
- [Background] Fukuoka M, Wu YL, Thongprasert S, Sunpaweravong P, Leong SS, Sriuranpong V, Chao TY, Nakagawa K, Chu DT, Saijo N, Duffield EL, Rukazenkov Y, Speake G, Jiang H, Armour AA, To KF, Yang JC, Mok TS. Biomarker analyses and final overall survival results from a phase III, randomized, open-label, first-line study of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer in Asia (IPASS). J Clin Oncol. 2011 Jul 20;29(21):2866-74. doi: 10.1200/JCO.2010.33.4235. Epub 2011 Jun 13. PMID 21670455
- [Background] Horgan AM, Bradbury PA, Amir E, Ng R, Douillard JY, Kim ES, Shepherd FA, Leighl NB. An economic analysis of the INTEREST trial, a randomized trial of docetaxel versus gefitinib as second-/third-line therapy in advanced non-small-cell lung cancer. Ann Oncol. 2011 Aug;22(8):1805-11. doi: 10.1093/annonc/mdq682. Epub 2011 Jan 27. PMID 21273345
- [Background] Douillard JY, Shepherd FA, Hirsh V, Mok T, Socinski MA, Gervais R, Liao ML, Bischoff H, Reck M, Sellers MV, Watkins CL, Speake G, Armour AA, Kim ES. Molecular predictors of outcome with gefitinib and docetaxel in previously treated non-small-cell lung cancer: data from the randomized phase III INTEREST trial. J Clin Oncol. 2010 Feb 10;28(5):744-52. doi: 10.1200/JCO.2009.24.3030. Epub 2009 Dec 28. PMID 20038723
- [Background] Kim ES, Hirsh V, Mok T, Socinski MA, Gervais R, Wu YL, Li LY, Watkins CL, Sellers MV, Lowe ES, Sun Y, Liao ML, Osterlind K, Reck M, Armour AA, Shepherd FA, Lippman SM, Douillard JY. Gefitinib versus docetaxel in previously treated non-small-cell lung cancer (INTEREST): a randomised phase III trial. Lancet. 2008 Nov 22;372(9652):1809-18. doi: 10.1016/S0140-6736(08)61758-4. PMID 19027483
- [Background] Lee DH, Park K, Kim JH, Lee JS, Shin SW, Kang JH, Ahn MJ, Ahn JS, Suh C, Kim SW. Randomized Phase III trial of gefitinib versus docetaxel in non-small cell lung cancer patients who have previously received platinum-based chemotherapy. Clin Cancer Res. 2010 Feb 15;16(4):1307-14. doi: 10.1158/1078-0432.CCR-09-1903. Epub 2010 Feb 9. PMID 20145166
- [Background] Maruyama R, Nishiwaki Y, Tamura T, Yamamoto N, Tsuboi M, Nakagawa K, Shinkai T, Negoro S, Imamura F, Eguchi K, Takeda K, Inoue A, Tomii K, Harada M, Masuda N, Jiang H, Itoh Y, Ichinose Y, Saijo N, Fukuoka M. Phase III study, V-15-32, of gefitinib versus docetaxel in previously treated Japanese patients with non-small-cell lung cancer. J Clin Oncol. 2008 Sep 10;26(26):4244-52. doi: 10.1200/JCO.2007.15.0185. PMID 18779611
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771
- [Derived] Marabese M, Ganzinelli M, Garassino MC, Shepherd FA, Piva S, Caiola E, Macerelli M, Bettini A, Lauricella C, Floriani I, Farina G, Longo F, Bonomi L, Fabbri MA, Veronese S, Marsoni S, Broggini M, Rulli E. KRAS mutations affect prognosis of non-small-cell lung cancer patients treated with first-line platinum containing chemotherapy. Oncotarget. 2015 Oct 20;6(32):34014-22. doi: 10.18632/oncotarget.5607. PMID 26416458
- [Derived] Rulli E, Marabese M, Torri V, Farina G, Veronese S, Bettini A, Longo F, Moscetti L, Ganzinelli M, Lauricella C, Copreni E, Labianca R, Martelli O, Marsoni S, Broggini M, Garassino MC; TAILOR trialists. Value of KRAS as prognostic or predictive marker in NSCLC: results from the TAILOR trial. Ann Oncol. 2015 Oct;26(10):2079-84. doi: 10.1093/annonc/mdv318. Epub 2015 Jul 24. PMID 26209642
- [Derived] Garassino MC, Martelli O, Broggini M, Farina G, Veronese S, Rulli E, Bianchi F, Bettini A, Longo F, Moscetti L, Tomirotti M, Marabese M, Ganzinelli M, Lauricella C, Labianca R, Floriani I, Giaccone G, Torri V, Scanni A, Marsoni S; TAILOR trialists. Erlotinib versus docetaxel as second-line treatment of patients with advanced non-small-cell lung cancer and wild-type EGFR tumours (TAILOR): a randomised controlled trial. Lancet Oncol. 2013 Sep;14(10):981-8. doi: 10.1016/S1470-2045(13)70310-3. Epub 2013 Jul 22. PMID 23883922
- [Derived] Farina G, Longo F, Martelli O, Pavese I, Mancuso A, Moscetti L, Labianca R, Bertolini A, Cortesi E, Farris A, Fagnani D, Locatelli MC, Valmadre G, Ardizzoia A, Tomirotti M, Rulli E, Garassino MC, Scanni A. Rationale for treatment and study design of tailor: a randomized phase III trial of second-line erlotinib versus docetaxel in the treatment of patients affected by advanced non-small-cell lung cancer with the absence of epidermal growth factor receptor mutations. Clin Lung Cancer. 2011 Mar;12(2):138-41. doi: 10.1016/j.cllc.2011.03.008. Epub 2011 Apr 11. PMID 21550561